CLINICAL TRIAL: NCT04644211
Title: A Phase 2 Study Of Ruxolitinib In Low-Risk Essential Thrombocythemia And Polycythemia Vera With Significant Symptom Burden
Brief Title: Ruxolitinib in Thrombocythemia and Polycythemia Vera
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Principal Investigator, Gabriela Hobbs, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20-364
Record Dates: First submitted 2020-11-10; First posted 2020-11-25 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Essential Thrombocythemia; Polycythemia Vera
Keywords: Essential Thrombocythemia; Polycythemia Vera; Sympton Burden
MeSH Terms: conditions — Thrombocythemia, Essential; Polycythemia Vera | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ruxolitinib Stage 1 (Experimental): In stage 1, participants will be divided into two cohorts:
  * Very low, Low, and Intermediate-risk ETpatients with significant symptom burden and Low-risk PV patients with significant symptom burden
  * Study cycles are 28 days long, participants in both cohorts will receive:
    * Ruxolitinib 2x daily for 6 study cycles.
  Interventions: Drug: Ruxolitinib
- Ruxolitinib Stage 2 (Experimental): Stage 2 will commence based on 3 or more participants in Stage 1 showing a predetermined positive response to Ruxolitinib.
  In stage 2, participants will be divided into two cohorts:
  * Very low, Low, and Intermediate-risk ET patients with significant symptom burden and Low-risk PV patients with significant symptom burden
  * Study cycles are 28 days long, participants in both cohorts will receive:
    * Ruxolitinib 2x daily for 6 study cycles.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Pill taken by mouth.
  Other Names: Jakafi

SUMMARY:
This research is being done to see if the drug ruxolitinib is effective in reducing the symptoms caused by low-risk essential thrombocythemia (ET) and polycythemia vera (PV).

- This research study involves the study drug Ruxolitinib.

DETAILED DESCRIPTION:
This is a multi-center, non-randomized, two-stage phase II clinical trial evaluating ruxolitinib in low-risk but symptomatic essential thrombocythemia (ET) and polycythemia vera (PV) patients. This research is being done to see if Ruxolitinib is effective in reducing the symptoms people with essential thrombocythemia (ET) and polycythemia vera (PV) are experiencing. Ruxolitinib is a type of drug that blocks the specific proteins that may be causing the symptoms people with essential thrombocythemia (ET) and polycythemia vera (PV are experiencing.

The research study procedures include screening for eligibility and study treatment, including evaluations and follow up visits.

- Participants will receive Ruxolitinib for approximately 6 months and if benefitting from it may continue to receive Ruxolitinib for as long as there is no unacceptable side effects or disease progression.

It is expected that about 60 people will take part in this research study.

The U.S. Food and Drug Administration (FDA) has approved Ruxolitinib for polycythemia vera (PV) but not for people with essential thrombocythemia (ET) and polycythemia vera (PV).

Incyte, a biopharmaceutical company, is supporting this research study by providing funding for the study, including the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been diagnosed with essential thrombocythemia or polycythemia vera by World Health Organization 2016 diagnostic criteria.
* Patients with essential thrombocythemia must be very low (no history of thrombosis, age <60, and no JAK2 mutation), low (no history of thrombosis, age <60, presence of JAK2 mutation), or intermediate risk (no history of thrombosis, age >60, no JAK2 mutation) by IPSET criteria. Patients with polycythemia vera must be low risk (no history of thrombosis and age <60) by NCCN guidelines.
* Patients with an MPN-SAF TSS (MPN-10) score >10 AND at least one individual feature >5 documented on a separate visit within 3 months prior to study registration, as documented in the clinical record or obtained by clinician. If not previously documented in the electronic medical record, participants must be blinded to purpose of MPN SAF TSS scoring for eligibility determination. Average daily MPN-SAF TSS (MPN-10) score must remain >10 with any individual feature >5 for the week-long baseline assessment prior to ruxolitinib initiation.
* Patients who have previously received or are receiving cytoreductive therapy (i.e. hydroxyurea, anagrelide, interferon) are eligible for the study if therapy was used for the indication of symptom control, or if therapy was used for pre-operative control of blood counts. If a subject is still receiving cytoreductive therapy at the time of screening and enrollment, there will be a wash-out period from prior cytoreductive therapy at least 7 days prior to ruxolitinib initiation.
* Age ≥18 years.
* ECOG performance status ≤2 (Karnofsky ≥60%)
* Participants must have adequate organ and marrow function as defined below:

  * leukocytes ≥3,000/mcL
  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * total bilirubin ≤ institutional upper limit of normal (ULN)
  * AST(SGOT)/ALT(SGPT) ≤3 × institutional ULN
  * creatinine ≤ institutional ULN OR glomerular filtration rate (GFR) ≥60 mL/min/1.73 m2 unless data exists supporting safe use at lower kidney function values, no lower than 30 mL/min/1.73 m2
* Participants with a prior or concurrent malignancy not receiving treatment for concurrent cancer diagnosis and/or prior concurrent malignancy within 5 years except for basal cell carcinoma or squamous cell carcinoma of the skin.
* For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* For participants with evidence of chronic human immunodeficiency virus (HIV) infection, they must be negative for HBV DNA, HCV RNA, or hepatitis B surface antigen (BsAg) on suppressive therapy, if indicated.
* Participants must be previously vaccinated with the Herpes Zoster (Shingles) vaccine or must be willing to start prophylactic Acyclovir 400 mg twice daily (BID) or suitable alternative for duration of treatment with ruxolitinib.
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants should be class 2B or better.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Essential thrombocythemia patients who are high risk by IPSET-R criteria (age > 60 with JAK2 V617F mutation and/or history of thrombosis).1 Polycythemia vera patients who are high risk by NCCN guidelines (age > 60 and/or history of thrombosis).
* Patients with >5% blasts on baseline marrow exam or at any other time in peripheral blood
* Participants who are receiving any other investigational agents.
* Participants with a history of splenectomy. Participants may still be eligible after discussion with and approval by the Overall PI, however.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ruxolitinib or excipients of ruxolitinib.
* Participants requiring any medications or substances that are strong inhibitors or 3A4 isozyme are ineligible. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the participant will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the participant is considering a new over-the-counter medicine or herbal product.
* Participants with uncontrolled intercurrent illness.
* Participants with inadequate liver or renal function at screening as evidenced by lab values not meeting criteria
* Participants with psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because ruxolitinib is a Class C agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ruxolitinib, breastfeeding should be discontinued if the mother is treated with ruxolitinib.
* The effects of ruxolitinib on the developing human fetus are unknown. Pregnant women and subjects of childbearing potential who are unwilling to take appropriate precautions to avoid becoming pregnant or fathering a child are ineligible. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of ruxolitinib administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2034-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who achieve >50% reduction from baseline to Myeloproliferative Neoplasm Symptom Assessment Total Symptom Score | baseline to 12 weeks
  Percentage of patients with >50% change in Myeloproliferative Neoplasm Symptom Assessment Total Symptom Score (MPN-SAF TSS), which has use in major clinical trials and as symptom assessment in all patients in clinical practice. Modeling has established baseline MPN-SAF TSS cut-off scores (total MPN-SAF TSS >20 or an individual component score >5) at which symptomatic treatment would be significantly beneficial

SECONDARY OUTCOMES:
Proportion of patients achieving complete hematologic rate at week 12 | Week 12
  Evaluate the efficacy of ruxolitinib in improving hematologic remission rates, as measured by International Working Group (IWG) working criteria ET: Platelet count ≤ 400 x 109/L, WBC count <10 x 109/L, and absence of leukoerythroblastosis PV: hematocrit <45% and WBC count <10 x 109/L
Proportion of patients achieving complete hematologic rate at 24 Weeks | Week 24
  Evaluate the efficacy of ruxolitinib in improving hematologic remission rates, as measured by International Working Group (IWG) working criteria ET: Platelet count ≤ 400 x 109/L, WBC count <10 x 109/L, and absence of leukoerythroblastosis PV: hematocrit <45% and WBC count <10 x 109/L
Best MPN-SAF TSS score | 12 Weeks
  Myeloproliferative Neoplasm Symptom Assessment Total Symptom Score (MPN-SAF TSS) for use in major clinical trials and as symptom assessment in all patients in clinical practice. Modeling has established baseline MPN-SAF TSS cut-off scores (total MPN-SAF TSS >20 or an individual component score >5) at which symptomatic treatment would be significantly beneficial. Scale title includes absence of symptom (0) and worst imaginable symptoms (10) per question, with minimum score 0 and maximum score 100. Higher scores indicate worse outcomes.
Best MPN-SAF TSS score | 24 Weeks
  Myeloproliferative Neoplasm Symptom Assessment Total Symptom Score (MPN-SAF TSS) for use in major clinical trials and as symptom assessment in all patients in clinical practice. Modeling has established baseline MPN-SAF TSS cut-off scores (total MPN-SAF TSS >20 or an individual component score >5) at which symptomatic treatment would be significantly beneficial. . Scale title includes absence of symptom (0) and worst imaginable symptoms (10) per question, with minimum score 0 and maximum score 100. Higher scores indicate worse outcomes.
Percentage of change in Spleen Volume | baseline to 12 weeks
  Spleen volume reduction will be measured as the change in percentage spleen volume from baseline at 12 weeks as measured by CT, or MRI in patients with medical contraindication to CT. Summary statistics will be used to describe changes in spleen volume. Volume will be calculated by a computer-assisted perimeter method based on Sorenson et al. Spleen and liver volume will be obtained by outlining the circumference of the organ and determining the volume using the validated technique of least squares
Number of Participants with Treatment Related Adverse Events as Assessed by CTCAE v 5.0 | All patients who initiate treatment with study drug up to 60 months
  descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for AE reporting

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Hobbs, MD, Principal Investigator — Massachusetts General Hospital
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth-Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General North Shore Cancer Center, Danvers, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation